CLINICAL TRIAL: NCT02684240
Title: A 14 Day Early Bactericidal Activity Study of Nitazoxanide for the Treatment of Tuberculosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1302013616
Record Dates: First submitted 2016-02-02; First posted 2016-02-17 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — nitazoxanide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nitazoxanide (Experimental): Participants with drug-sensitive tuberculous randomized to the NTZ arm will receive nitazoxanide 1000 mg po twice daily for 14 days. After this time point, participants will be switched to WHO standard tuberculosis therapy with isoniazid, rifampin, pyrazinamide and ethambutol.
  Interventions: Drug: Nitazoxanide
- Control (Other): Participants with drug-sensitive tuberculosis randomized to the standard therapy arm will receive WHO standard tuberculosis therapy involving isoniazid 300 mg po daily, rifampin 600 mg po daily, pyrazinamide 25 mg/kg po daily and ethambutol 15 mg/kg po daily.
  Interventions: Other: Control

INTERVENTIONS:
Drug: Nitazoxanide — nitazoxanide 1000 mg orally twice daily with food for 14 days
  Other Names: Nizonide; Alinia
  Arms: Nitazoxanide
Other: Control — The control arm will receive WHO standard therapy for tuberculosis with isoniazid, rifampin, pyrazinamide, and ethambutol
  Arms: Control

SUMMARY:
This research is being done to determine if Nitazoxanide (NTZ) will cause a significant decrease in the number of M. tuberculosis bacteria in sputum after 14 days of treatment. The study is being conducted at the GHESKIO Centers in Port au Prince Haiti

DETAILED DESCRIPTION:
This is a prospective randomized two-arm 14-day, early bactericidal activity study in treatment-naive, drug-susceptible patients with uncomplicated pulmonary tuberculosis (TB). The study will be conducted at the GHESKIO Centers in Port au Prince Haiti. Twenty patients will be randomized to receive NTZ 1 gram orally twice daily for 14 days. Ten patients will be randomized as positive controls to receive standard 4 drug tuberculosis therapy with isoniazid (H), rifampin (R), ethambutol (E), and pyrazinamide (PZA). Patients' sputum will be collected before and then every two days during 14 days of treatment, and the primary endpoint will be the change in the number of M. tuberculosis in patients' sputum. Our primary hypothesis is that NTZ will result in a significant decrease in the number of M. tuberculosis in sputum during14 days of treatment. The number of M. tuberculosis will be quantified by the time to positive (TTP) signal in hours in an automated liquid media culture system (BACTEC MGIT 960, Becton Dickinson).

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18 - 65
* Diagnosed with pulmonary tuberculosis via: sputum-microscopy smear-positive (2+ or 3+) within 14 days plus Sputum GeneXpert positive within 14 days plus Chest radiograph consistent with M. tuberculosis within 14 days
* TB treatment naïve at time of enrollment
* Bodyweight > 40kg
* Negative HIV test within 30 days
* Able to complete activities of daily living (ADLs)
* All participants must agree not to participate in a conception process (i.e. active attempt to become pregnant or to impregnate, donate sperm, in vitro fertilization)
* All female participants must agree to use barrier methods such as condoms as well as hormonal contraception for dual prophylaxis.
* Able to give informed consent and demonstrate understanding of this study and willingness to participate in this study
* Willing to be hospitalized for 2 weeks

Exclusion Criteria:

* Pregnancy
* Evidence of complications of M. tuberculosis such as hemoptysis or shortness of breath
* Extrapulmonary manifestations of M. tuberculosis
* History of prior active tuberculosis
* Evidence of rifampin resistance via GeneXpert
* Previous diagnosis of diabetes or suggestion of impaired glucose metabolism via random plasma glucose
* Previous diagnosis of HIV by any rapid HIV test or by ELISA
* Any of the following lab abnormalities: Creatinine > 1.5 times the ULN; Random glucose > 2 times the ULN; ALT, AST, or alkaline phosphatase > 2 times the ULN; Hemoglobin < 7.5 g/dL
* Any participant currently taking antimycobacterial therapy or within the past 30 days
* Any concomitant illness that could compromise patient safety in this trial such as renal failure, chronic liver disease or alcoholic dependency
* Enrolled in another clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-02; Primary Completion 2018-04-11 (Actual); Study Completion 2018-04-11 (Actual)

PRIMARY OUTCOMES:
time to positivity (TTP) | first 14 days of anti-tuberculosis therapy
  To assess the change in time in hours to positive (TTP) signal in an automated liquid media culture system (BACTEC MGIT 960, Becton Dickinson) in participants receiving NTZ over 14 days

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as determined by DAIDS toxicity tables | first 14 days of anti-tuberculosis therapy
  To assess the safety of 1000 mg twice daily dosing of NTZ in participants with drug-sensitive tuberculosis by grading each treatment-related adverse reaction according the DAIDS Toxicity tables (November 2014)
Maximum plasma concentration of NTZ | first 14 days of anti-tuberculosis therapy
  To assess the maximum plasma concentration of NTZ via collection of whole blood samples at hours 2, 4, 6 after ingestion of 1000 mg NTZ on day 5 and day 14 of the study
Most probable number of M tuberculosis in 1 ml of sputum | first 14 days of anti-tuberculosis therapy
  To quantify the number of M. tuberculosis (MTB) in sputum at baseline and at day 14 using most probable number (MPN) micro-plate assay with and without resuscitation factors added to media
First-line drug susceptibility (DST) of Mycobacterium tuberculosis via Mycobacterial Growth Indicator System (MGIT) | first 14 days of anti-tuberculosis therapy
  To test for first-line drug susceptibility (DST) of Mycobacterium tuberculosis to isoniazid, rifampin, pyrazinamide and ethambutol via MGIT
Quantification of change in urine metabolites and correlation with change in TTP | first 14 days of anti-tuberculosis therapy
  To quantify the change in urine metabolites by LC-MS technology and the correlation of this change with change in TTP.
Minimum plasma concentration of NTZ | first 14 days of anti-tuberculosis therapy
  To assess the minimum plasma concentration of NTZ via collection of whole blood samples at 30 minutes prior to ingestion of 1000 mg of NTZ on day 5 and day 14 of the study
Area under the curve of NTZ metabolites | first 14 days of anti-tuberculosis therapy
  To assess the area under the curve of NTZ metabolites (tizoxanide, tizoxanide glucuronide) via collection of whole blood samples at hour 2, 4, and 6 post-ingestion of 1000 mg of NTZ on day 5 and day 14
Sputum concentration of NTZ | first 14 days of anti-tuberculosis therapy
  To assess the sputum concentration of NTZ via collection of spot sputum samples 4 hours post-ingestion of 1000 mg NTZ on day 5 and day 14 of study
Change in Minimum inhibitory concentration (MIC) of NTZ against Tuberculosis over 14 days | first 14 days of anti-tuberculosis therapy
  To assess the MIC of NTZ against tuberculosis using microplate assay at baseline and again at day 14 to determine any change in the MIC over the course of treatment
Change in phylogeny of bacteria determined by sequencing of amplified 16S ribosomal DNA and/or metagenomic sequencing of bacterial DNA | first 14 days of anti-tuberculosis therapy
  Change in phylogeny of bacteria determined by sequencing of amplified 16S ribosomal DNA and/or metagenomic sequencing of bacterial DNA over the course of 14 days and correlation of this change with change in TTP.
Transcriptional signature of treatment response using whole blood transcriptional profiles | first 14 days of anti-tuberculosis therapy
  Determine the transcriptional signature of treatment response using whole blood transcriptional profiles obtained at baseline and day 14

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W Fitzgerald, MD, Principal Investigator — Weill Medical College of Cornell University; Carl Nathan, MD, Study Chair — Weill Medical College of Cornell University; Jean William Pape, MD, Study Chair — Groupe Haitien d'Etude du Sarcome de Kaposi et des Infections Opportunistes (GHESKIO)
Locations (1):
- Les Centres GHESKIO, Port-au-Prince, Haiti

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared once the trial is complete. Data is currently being analyzed.

REFERENCES:
- [Background] de Carvalho LP, Lin G, Jiang X, Nathan C. Nitazoxanide kills replicating and nonreplicating Mycobacterium tuberculosis and evades resistance. J Med Chem. 2009 Oct 8;52(19):5789-92. doi: 10.1021/jm9010719. PMID 19736929
- [Background] Stockis A, De Bruyn S, Gengler C, Rosillon D. Nitazoxanide pharmacokinetics and tolerability in man during 7 days dosing with 0.5 g and 1 g b.i.d. Int J Clin Pharmacol Ther. 2002 May;40(5):221-7. doi: 10.5414/cpp40221. PMID 12051574
- [Background] Shigyo K, Ocheretina O, Merveille YM, Johnson WD, Pape JW, Nathan CF, Fitzgerald DW. Efficacy of nitazoxanide against clinical isolates of Mycobacterium tuberculosis. Antimicrob Agents Chemother. 2013 Jun;57(6):2834-7. doi: 10.1128/AAC.02542-12. Epub 2013 Mar 18. PMID 23507275
- [Result] Walsh KF, McAulay K, Lee MH, Vilbrun SC, Mathurin L, Jean Francois D, Zimmerman M, Kaya F, Zhang N, Saito K, Ocheretina O, Savic R, Dartois V, Johnson WD, Pape JW, Nathan C, Fitzgerald DW. Early Bactericidal Activity Trial of Nitazoxanide for Pulmonary Tuberculosis. Antimicrob Agents Chemother. 2020 Apr 21;64(5):e01956-19. doi: 10.1128/AAC.01956-19. Print 2020 Apr 21. PMID 32071052
- [Derived] Wipperman MF, Bhattarai SK, Vorkas CK, Maringati VS, Taur Y, Mathurin L, McAulay K, Vilbrun SC, Francois D, Bean J, Walsh KF, Nathan C, Fitzgerald DW, Glickman MS, Bucci V. Gastrointestinal microbiota composition predicts peripheral inflammatory state during treatment of human tuberculosis. Nat Commun. 2021 Feb 18;12(1):1141. doi: 10.1038/s41467-021-21475-y. PMID 33602926